CLINICAL TRIAL: NCT01362790
Title: A Pilot/ Phase 2 Study of Pentostatin Plus Cyclophosphamide Immune Depletion to Decrease Immunogenicity of SS1P in Patients With Mesothelioma, Lung Cancer or Pancreatic Cancer
Brief Title: SS1P and Pentostatin Plus Cyclophosphamide for Mesothelioma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Raffit Hassan, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 110160; 11-C-0160
Record Dates: First submitted 2011-05-27; First posted 2011-05-30 (Estimated); Results first posted 2019-06-06 (Actual); Last update posted 2019-06-06 (Actual); Status verified 2019-06

CONDITIONS: Mesothelioma; Adenocarcinoma of Lung; Pancreatic Neoplasms
Keywords: Immune Therapy; Immunotoxin; T-Cell Depletion; Mesothelioma
MeSH Terms: conditions — Mesothelioma; Adenocarcinoma of Lung; Pancreatic Neoplasms | interventions — Pentostatin; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Mesothelioma Pilot Phase Regimen A (Experimental): Drug: Pentostatin Regimen A: Cycle 1: 4 mg/m^2 on days 1, 5 and 9 of 30 day cycle Cycles 2-4: 4 mg/m^2 on day 1 of 21 day cycle
  Other Names:
  • Nipent Drug: Cyclophosphamide Regimen A:Cycle 1: 200 mg/day on days 1-12 of 30 day cycle Cycles 2-4: 200 mg/day on days 1-4 of 21 day cycle
  Other Names:
  • Cytoxan Drug: SS1 (dsFv)PE38 Regimen A: Cycle 1: 35 mcg/kg days 10, 12, and 14. Cycles 2-4: Days 2, 4, and 6, for a maximum of six treatment cycles.
  Interventions: Drug: Pentostatin; Drug: Cyclophosphamide; Biological: SS1(dsFv)PE38 - lot 073I0809; Biological: SS1(dsFv)PE38 - lot FIL129J01
- Mesothelioma Pilot Phase Regimen B (Experimental): Drug: Pentostatin Regimen B: Cycle 1: 4 mg/m^2 or 2 mg/m^2 on days 1, 5, 9, 13 and 17 of 38 day cycle Cycles 2-6: 4 mg/m^2 on days 1 and 5 of 25 day cycle Regimen B: Cycle 1: 4 mg/m^2 on days 1, 5, 9, 13 and 17 of 38 day cycle Cycles 2-6: 4 mg/m^2 on days 1 and 5 of 25 day cycle
  Other Names:
  • Nipent Drug: Cyclophosphamide Regimen B:Cycle 1: 200 mg/day on days 1-20 of 38 day cycle Cycles 2-4: 200 mg/day on days 1-8 of 25 day cycle
  Other Names:
  • Cytoxan Drug: SS1 (dsFv)PE38 Regimen B: Cycle 1: 35mcg/kg days 18, 20, and 22. Cycles 2-4: (Days 6, 8, and 10), for a maximum of six treatment cycles.
  Interventions: Drug: Pentostatin; Drug: Cyclophosphamide; Biological: SS1(dsFv)PE38 - lot 073I0809; Biological: SS1(dsFv)PE38 - lot FIL129J01
- Phase 2 Peritoneal Mesothelioma Pilot Expansion Phase (Experimental): Drug: Pentostatin Regimen B: Cycle 1: 4 mg/m^2 or 2 mg/m^2 on days 1, 5 and 9 of 38 day cycle Cycles 2-6: 4 mg/m^2 on day 1 and 5 of 25 day cycle
  Other Names:
  • Nipent Drug: Cyclophosphamide Regimen B:Cycle 1: 200 mg/day on days 1-20 of 38 day cycle Cycles 2-4: 200 mg/day on days 1-8 of 25 day cycle
  Other Names:
  • Cytoxan Drug: SS1(dsFv)PE38 Regimen B: Cycle 1: 35 mcg/kg or 25 mcg/kg days 18, 20 and 22. Cycles 2-4: Days 6, 8, and 10, for a maximum of six treatment cycles.
  Interventions: Drug: Pentostatin; Drug: Cyclophosphamide; Biological: SS1(dsFv)PE38 - lot 073I0809; Biological: SS1(dsFv)PE38 - lot FIL129J01
- Phase 2 Pleural Mesothelioma Pilot Expansion Phase (Experimental): Drug: Pentostatin Regimen A: Cycle 1: 4 mg/m^2 on days 1, 5 and 9 of 30 day cycle Cycles 2-4: 4 mg/m^2 on day 1 of 21 day cycle
  Other Names:
  • Nipent Drug: Cyclophosphamide Regimen A:Cycle 1: 200 mg/day on days 1-12 of 30 day cycle Cycles 2-4: 200 mg/day on days 1-4 of 21 day cycle
  Other Names:
  • Cytoxan Drug: SS1(dsFv)PE38 Regimen A: Cycle 1: 35 mcg/kg or 25 mcg/kg days 10, 12 and 14. Cycles 2-4: Days 2, 4, and 6, for a maximum of six treatment cycles.
  Interventions: Drug: Pentostatin; Drug: Cyclophosphamide; Biological: SS1(dsFv)PE38 - lot 073I0809; Biological: SS1(dsFv)PE38 - lot FIL129J01
- Mesothelioma Positive Ca Dose De-escalation Pilot Regimen A (Experimental): Drug: Pentostatin Regimen A: Cycle 1: 4 mg/m^2 on days 1, 5 and 9 of 30 day cycle Cycles 2-4: 4 mg/m^2 on day 1 of 21 day cycle
  Other Names:
  • Nipent Drug: Cyclophosphamide Regimen A:Cycle 1: 200 mg/day on days 1-12 of 30 day cycle Cycles 2-4: 200 mg/day on days 1-4 of 21 day cycle
  Other Names:
  • Cytoxan Drug: SS1(dsFv)PE38 Regimen A: Cycle 1: 35 mcg/kg or 25 mcg/kg days 10, 12 and 14. Cycles 2-4: Days 2, 4, and 6, for a maximum of six treatment cycles.
  Interventions: Drug: Pentostatin; Drug: Cyclophosphamide; Biological: SS1(dsFv)PE38 - lot 073I0809; Biological: SS1(dsFv)PE38 - lot FIL129J01
- Phase 2 Pancreatic Adenocarcinoma Pilot Phase Regimen A (Experimental): Drug: Pentostatin Regimen A: Cycle 1: 4 mg/m^2 on days 1, 5 and 9 of 30 day cycle Cycles 2-4: 4 mg/m^2 on day 1 of 21 day cycle
  Other Names:
  • Nipent Drug: Cyclophosphamide Regimen A:Cycle 1: 200 mg/day on days 1-12 of 30 day cycle Cycles 2-4: 200 mg/day on days 1-4 of 21 day cycle
  Other Names:
  • Cytoxan Drug: SS1(dsFv)PE38 Regimen A: Cycle 1: 35 mcg/kg or 25 mcg/kg days 10, 12 and 14. Cycles 2-4: Days 2, 4, and 6, for a maximum of six treatment cycles.
  Interventions: Drug: Pentostatin; Drug: Cyclophosphamide; Biological: SS1(dsFv)PE38 - lot 073I0809; Biological: SS1(dsFv)PE38 - lot FIL129J01
- Phase 2 Lung Adenocarcinoma Pilot Expansion Phase Regimen A (Experimental): Drug: Pentostatin Regimen A: Cycle 1: 4 mg/m^2 on days 1, 5 and 9 of 30 day cycle Cycles 2-4: 4 mg/m^2 on day 1 of 21 day cycle
  Other Names:
  • Nipent Drug: Cyclophosphamide Regimen A:Cycle 1: 200 mg/day on days 1-12 of 30 day cycle Cycles 2-4: 200 mg/day on days 1-4 of 21 day cycle
  Other Names:
  • Cytoxan Drug: SS1(dsFv)PE38 Regimen A: Cycle 1: 35 mcg/kg or 25 mcg/kg days 10, 12 and 14. Cycles 2-4: Days 2, 4, and 6, for a maximum of six treatment cycles.
  Interventions: Drug: Pentostatin; Drug: Cyclophosphamide; Biological: SS1(dsFv)PE38 - lot 073I0809; Biological: SS1(dsFv)PE38 - lot FIL129J01

INTERVENTIONS:
Drug: Pentostatin — Regimen A: Cycle 1: 4 mg/m^2 on days 1, 5 and 9 of 30 day cycle Cycles 2-4: 4 mg/m^2 on day 1 of 21 day cycle Regimen B: Cycle 1: 4 mg/m^2 or 2 mg/m^2 on days 1, 5, 9, 13 and 17 of 38 day cycle Cycles 2-6: 4 mg/m^2 on days 1 and 5 of 25 day cycle
  Other Names: Nipent
Drug: Cyclophosphamide — Regimen A:Cycle 1: 200 mg/day on days 1-12 of 30 day cycle Cycles 2-4: 200 mg/day on days 1-4 of 21 day cycle Regimen B:Cycle 1: 200 mg/day on days 1-20 of 38 day cycle Cycles 2-4: 200 mg/day on days 1-8 of 25 day cycle
  Other Names: Cytoxan
Biological: SS1(dsFv)PE38 - lot 073I0809 — Regimen A: Cycle 1: Cycle 1: 35mcg/kg days 10, 12 and 14 Cycles 2-4: Days 2, 4 and 6, for a maximum of six treatment cycles Regimen B: Cycle 1: 35mcg/kg days 18, 20 and 22 Cycles 2-4: (Days 6, 8 and 10), for a maximum of six treatment cycles
Biological: SS1(dsFv)PE38 - lot FIL129J01 — Regimen A:
  Cycle 1: Cycle 1:35mcg/kg or 25 mcg/kg days 10, 12 and 14 Cycles 2-4: Days 2, 4 and 6, for a maximum of six treatment cycles

SUMMARY:
Background:

* Malignant mesothelioma is a form of cancer that develops on the protective lining that covers the body's internal organs. It most often occurs on the lining of the lungs and chest wall or the lining of the abdomen. There is no known cure for malignant mesothelioma, so researchers are searching for new ways to treat it.
* Mesothelin is a protein that is found in mesothelioma and other types of cancer cells. An experimental cancer drug called SS1P is designed to attack cells that have mesothelin while leaving healthy cells alone. Researchers want to test how effective SS1P is when it is given with pentostatin and cyclophosphamide. These drugs help suppress the immune system and may make the SS1P more effective.

Objectives:

- To study the effectiveness of SS1P plus two drugs that suppress the immune system to treat malignant mesothelioma.

Eligibility:

- Individuals at least 18 years of age who have malignant mesothelioma in the chest or abdomen.

Design:

* Participants will be screened with a physical exam, medical history, and blood tests. They will also have imaging studies.
* The first treatment cycle will last 30 days. Up to three 21-day cycles of treatment will follow.
* In the first cycle, participants will have pentostatin on days 1, 5, and 9. They will have cyclophosphamide on days 1 through 12. They will have SS1P on days 10, 12, and 14.
* On the next three cycles, participants will have pentostatin on day 1.They will have cyclophosphamide on days 1 through 4. They will have SS1P on days 2, 4, and 6.
* Participants will have frequent blood tests and other studies. They will receive all four cycles of treatment as long as there are no severe side effects.
* Participants will have regular followup visits as directed by the study doctors.

DETAILED DESCRIPTION:
BACKGROUND:

Mesothelin is a cell surface glycoprotein present on normal mesothelial cells that is highly expressed in many human cancers including mesothelioma, lung and pancreatic adenocarcinoma. SS1 (dsFv) PE38 is a recombinant anti-mesothelin immunotoxin that has undergone phase I testing and has been evaluated in combination with pemetrexed and cisplatin for treatment of malignant pleural mesothelioma. SS1 (dsFv)PE38 is highly immunogenic and the majority of patients develop antibodies to it at end of one cycle. Pre-clinical studies demonstrate that SS1(dsFv)PE38 may be administered multiple times in combination with an immune-depleting regimen consisting of pentostatin and cyclophosphamide.

OBJECTIVES:

Mesothelioma Pilot Objective

-To assess the safety, tolerability, and feasibility of a conditioning regimen of pentostatin

and cyclophosphamide in combination with SS1(dsFv)PE38

-To monitor antibody formation to SS1(dsFv)PE38 and to assess the impact of the conditioning regimen on the formation of these antibodies

Mesothelioma Positive Cancers Dose De-escalation Pilot Objective

-To determine the safety profile and recommended phase 2 dose of SS1P (dsFv)PE38 in

drug lot FIL129J01 using dosing regimen A in patients with mesothelioma, lung and pancreatic adenocarcinoma

Phase 2 and Lung and Pancreatic Adenocarcinoma Expansion Pilot Objective

-To evaluate objective tumor response in subjects with pleural mesothelioma, peritoneal

mesothelioma, lung and pancreatic adenocarcinoma using Regimen A

ELIGIBILITY:

* Patients with one of the following histologically confirmed malignancies:

  * malignant pleural or peritoneal mesothelioma with epithelial or biphasic tumors having less than a 50% sarcomatoid component who have previously been treated on at least one platinum-containing chemotherapy regimen with progressive disease documented prior to study entry
  * advanced (Stage IIIB/IV) lung adenocarcinoma who have had at least one prior chemotherapy for advanced disease. Patients who received an approved targeted therapy as first-line treatment should have also received chemotherapy prior to study entry.
  * recurrent, locally advanced unresectable or metastatic adenocarcinoma of the pancreas.
* Measurable disease by modified Response Evaluation Criteria in Solid Tumors (RECIST) criteria for pleural mesothelioma or by RECIST criteria for peritoneal mesothelioma, lung adenocarcinoma and pancreatic adenocarcinoma

  * Adequate renal, hepatic and hematopoietic function
  * No major surgery, radiotherapy, chemotherapy or biologic therapy within 28 days of therapy

DESIGN:

-During the mesothelioma pilot phase of this study, the first eleven mesothelioma patients

enrolled in this study received a conditioning regimen of pentostatin on days 1, 5 and 9 of the first cycle and day 1 of subsequent cycles in combination with cyclophosphamide on days 1 through 12 of the first cycle and days 1 through 4 of subsequent cycles (Regimen A) while the next 8 mesothelioma patients received conditioning regimen of pentostatin on days 1, 5, 9, 13 and 17 of the first cycle and day 1 and 5 of subsequent cycles in combination with cyclophosphamide on days 1 through 20 of the first cycle and days 1 through 8 of subsequent cycles (Regimen B). SS1P was administered every other day for six days (3 doses) beginning on the day after the last pentostatin dose in each cycle for both regimens.

* In the mesothelin positive cancers dose de-escalation pilot study, a maximum of 12 patients with mesothelioma or lung or pancreatic adenocarcinoma will be enrolled in a 3+3 design to test up to 2 decreasing dose levels of SS1P administered in combination with cyclophosphamide and pentostatin on the Regimen A schedule for safety.
* In the phase 2 mesothelioma and pancreatic and lung adenocarcinoma pilot expansion portions of the study, a two-stage Minimax phase II trial design will be used to enroll up to 16 evaluable subjects with pleural mesothelioma (cohort 1), up to 10 evaluable subjects with peritoneal mesothelioma (cohort 2), up to 10 patients with lung adenocarcinoma (cohort 3)and up to 10 evaluable subjects with pancreatic adenocarcinoma (cohort 4) who will receive treatment on Regimen A.
* Treatment cycles will be repeated for up to four cycles if patients do not develop neutralizing antibodies, which will be assessed by a biological assay 14 and 20 days (+/- 2 days) following the first dose of SS1P in each cycle (corresponding to Days 24 and 30 of Cycle 1, and Days 16 and 22 of Cycles 2 through 4)
* Toxicity will be assessed by the Cancer Therapy Evaluation Program (CTEP) Version 4.0 of Common Terminology Criteria in Adverse Events (CTCAE)
* Tumor response assessments will be performed at the end of 2 cycles and at the end of treatment
* Tumor biopsies will be performed before treatment, after 2 cycles, and after the last cycle or at follow-up.

ELIGIBILITY:
* INCLUSION CRITERIA: Mesothelioma Cohorts (Cohorts 1 and 2 Only)
* Subjects must have histologically confirmed epithelial or biphasic mesothelioma not amenable to potentially curative surgical resection. However, patients with biphasic tumors that have a less than or equal to 50% sarcomatoid component will be excluded. The diagnosis will be confirmed by the Laboratory of Pathology / Center for Cancer Research (CCR) / National Cancer Institute (NCI).
* Patients must have had at least one prior chemotherapy regimen, with the Food and Drug Administration (FDA) approved regimen of a platinum-based therapy in combination with pemetrexed being preferred unless there was a specific contraindication for an individual patient. There is no limit to the number of prior chemotherapy regimens received.
* Total Bilirubin less than or equal to 1.5 X institutional upper limit of normal (ULN)

INCLUSION CRITERIA: Lung Adenocarcinoma Cohort (Cohort 3) Only

* Subjects must have histologically confirmed advanced (Stage IIIB/IV) lung adenocarcinoma. The diagnosis will be confirmed by the Laboratory of Pathology/CCR/NCI.
* Patients must have had at least one prior therapy for advanced disease [platinum containing chemotherapy or one of the approved targeted therapies (an approved estimated glomerular filtration rate (EGFR) tyrosine kinase inhibitor (TKI) for EGFR mutant tumors or crizotinib and ceritinib for ALK translocated tumors)]. There is no limit to the number of prior chemotherapy regimens received.
* Mesothelin expression in at least 5% of cells as assessed in archival tumor tissue samples, determined by the immunohistochemistry (IHC) assay performed at Laboratory of Pathology / CCR / NCI. Archival samples must be available for eligibility.
* Total Bilirubin less than or equal to 1.5 X institutional upper limit of normal (ULN)

INCLUSION CRITERIA: Pancreatic Cancer Cohort (Cohort 4) Only

* Subjects with recurrent, locally advanced unresectable or metastatic adenocarcinoma of the pancreas. The diagnosis will be confirmed by the Laboratory of Pathology/CCR/NCI.
* Patients must have had at least one prior chemotherapy for advanced disease. There is no limit to the number of prior chemotherapy regimens received.
* Total Bilirubin less than or equal to 2 X institutional upper limit of normal (ULN)

INCLUSION CRITERIA: All Subjects

* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as >20 mm with conventional techniques or as >10 mm with spiral CT scan. See Section 11 for the evaluation of measurable disease.
* Patients must not have had major surgery, radiation therapy, chemotherapy, biologic therapy (including any investigational agents), or hormonal therapy (other than replacement), within 4 weeks prior to entering the study and must have evidence of stable or progressive disease to be eligible.
* Age greater than or equal to 18 years. Since the study diseases are extremely rare in children they are excluded from this study.
* Performance status (Eastern Cooperative Oncology Group (ECOG)) less than or equal to 1
* Patients must have adequate organ and marrow function (as defined below).

  * leukocytes less than or equal to 3,000/mm^3
  * absolute neutrophil count less than or equal to 1,500/mm^3
  * hemoglobin less than or equal to 9 g/dL
  * platelets less than or equal to 90,000/ mm^3
  * total bilirubin See guidelines for individual cohorts in sections 3.1.1.3, 3.1.2.4 and 3.1.3.3
  * Aspartate aminotransferase (AST)(serum glutamic oxaloacetic transaminase (SGOT))/alanine aminotransferase (ALT)(serum glutamic-pyruvic transaminase (SGPT)) less than or equal to 3 X institutional upper limit of normal (ULN) (5x if liver function test (LFT) elevations due to liver metastases)
  * creatinine less than or equal to 1.5 X institutional ULN

OR

--creatinine clearance greater than or equal to 45 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal, obtained through calculated or measured Creatinine Clearance

Patients may be transfused to obtain a hemoglobin of less than or equal to 9 g/Dl.

* The effects of SS1(dsFv)PE38, pentostatin, and cyclophosphamide on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (barrier method of birth control; abstinence) for the duration of study therapy and for 3 months after the last dose of therapy. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately. While hormonal methods of birth control are effective, we ask that female patients who are participating in the study cease hormonal forms of birth control, as these methods of birth control (birth control pills, injections, or implants) may affect the study drug. Patients must be off hormonal forms of birth control for at least 4 weeks prior to initiating the study.
* Ability to comply with intravenous administration schedule, and the ability to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA: (All Subjects)

* Patients with symptomatic brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events. However, patients who have had treatment for their brain metastases and whose brain metastatic disease status has remained stable for at least 4-6 weeks without steroids may be enrolled at the discretion of the principal investigator.
* Uncontrolled medical illness including, but not limited to, ongoing or uncontrolled, symptomatic congestive heart failure (American Heart Association (AHA) Class II or worse), uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Human immunodeficiency virus (HIV) positive patients will be excluded due to a theoretical concern that the degree of immune suppression associated with the treatment may result in progression of HIV infection.
* Patients with Hepatitis B and C will be excluded.
* Serum neutralization antibody assay shows greater than or equal to 75% neutralization of the SS1 (dsFv) PE38 activity at 200 ng/ml.
* Patients may not be receiving any other investigational agents.
* History of another invasive malignancy in the last two years. Adequately treated noninvasive, non-melanoma skin cancers as well as in situ carcinoma of the cervix will be allowed.
* Prior treatment with drugs of the immunotoxin class.
* Patients with tumor amenable to potentially curative therapy as assessed by the investigator.
* Pregnant women are excluded from this study because SS1(dsFv)PE38, pentostatin, and cyclophosphamide have the potential for teratogenic or abortifacient effects. The agents in the trial may also potentially be secreted in milk and therefore breastfeeding women should be excluded. Because of the potential of teratogenic or abortifacient effects women of childbearing potential and men must agree to use adequate contraception (barrier methods) before, during the study and for a period of 3 months after the last dose of the investigational agent.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to SS1(dsFv)PE38.

INCLUSION CRITERIA: WOMEN AND MINORITIES

-Both men and women and members of all races and ethnic groups are eligible for this trial. Every effort will be made to recruit women and minorities in this study.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2011-05-11 (Actual); Primary Completion 2016-08-03 (Actual); Study Completion 2017-08-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raffit Hassan, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hassan R, Bullock S, Premkumar A, Kreitman RJ, Kindler H, Willingham MC, Pastan I. Phase I study of SS1P, a recombinant anti-mesothelin immunotoxin given as a bolus I.V. infusion to patients with mesothelin-expressing mesothelioma, ovarian, and pancreatic cancers. Clin Cancer Res. 2007 Sep 1;13(17):5144-9. doi: 10.1158/1078-0432.CCR-07-0869. PMID 17785569
- [Background] Kay NE, Geyer SM, Call TG, Shanafelt TD, Zent CS, Jelinek DF, Tschumper R, Bone ND, Dewald GW, Lin TS, Heerema NA, Smith L, Grever MR, Byrd JC. Combination chemoimmunotherapy with pentostatin, cyclophosphamide, and rituximab shows significant clinical activity with low accompanying toxicity in previously untreated B chronic lymphocytic leukemia. Blood. 2007 Jan 15;109(2):405-11. doi: 10.1182/blood-2006-07-033274. Epub 2006 Sep 28. PMID 17008537
- [Background] Zhang Y, Xiang L, Hassan R, Paik CH, Carrasquillo JA, Jang BS, Le N, Ho M, Pastan I. Synergistic antitumor activity of taxol and immunotoxin SS1P in tumor-bearing mice. Clin Cancer Res. 2006 Aug 1;12(15):4695-701. doi: 10.1158/1078-0432.CCR-06-0346. PMID 16899620
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2011-C-0160.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 55 participants were enrolled. No data was collected for 10/55 participants who were screened for neutralizing antibodies and were positive, thus not enrolled into a Group /Arm, nor treated. 45/55 participants were treated on this study.
Groups:
- Phase 2 Peritoneal Mesothelioma Pilot Expansion Phase; Phase 2 Pleural Mesothelioma Pilot Expansion Phase; Phase 2 Pancreatic Adenocarcinoma Pilot Phase Regimen A; Phase 2 Lung Adenocarcinoma Pilot Expansion Phase Regimen A: Drug: Pentostatin Regimen A: Cycle 1: 4 mg/m^2 on days 1, 5 and 9 of 30 day cycle Cycles 2-4: 4 mg/m^2 on day 1 of 21 day cycle
  Other Names:
  • Nipent Drug: Cyclophosphamide Regimen A:Cycle 1: 200 mg/day on days 1-12 of 30 day cycle Cycles 2-4: 200 mg/day on days 1-4 of 21 day cycle
  Other Names:
  • Cytoxan Drug: SS1(dsFv)PE38 Regimen A: Cycle 1: 35 mcg/kg or 25 mcg/kg days 10, 12 and 14. Cycles 2-4: Days 2, 4, and 6, for a maximum of six treatment cycles.
- Mesothelioma Positive Ca Dose De-escalation Pilot Regimen A: Drug: Pentostatin Regimen A: Cycle 1: 4 mg/m^2 on days 1, 5 and 9 of 30 day cycle Cycles 2-4: 4 mg/m^2 on day 1 of 21 day cycle
  Other Names:
  • Nipent Drug: Cyclophosphamide Regimen A:Cycle 1: 200 mg/day on days 1-12 of 30 day cycle Cycles 2-4: 200 mg/day on days 1-4 of 21 day cycle
  Other Names:
  • Cytoxan Drug: SS1(dsFv)PE38 Regimen A: Cycle 1: 35 mcg/kg or 25 mcg/kg days 10, 12 and 14. Cycles 2-4: Days 2, 4, and 6, for a maximum of six treatment cycles.
  During Phase 2 SS1P was administered from 2 different Lots at 35mcg/kg (Lot F1L129J01 and Lot07310809). It was discovered that Lot F1L129J01 was more potent than Lot 07310809, therefore, a dose de-escalation was done for 8 participants who received that Lot to determine the MTD specific to the Lot.
Period: Pilot Phase & Phase 2
Arm/Group | Mesothelioma Pilot Phase Regimen A | Mesothelioma Pilot Phase Regimen B | Phase 2 Peritoneal Mesothelioma Pilot Expansion Phase | Phase 2 Pleural Mesothelioma Pilot Expansion Phase | Mesothelioma Positive Ca Dose De-escalation Pilot Regimen A | Phase 2 Pancreatic Adenocarcinoma Pilot Phase Regimen A | Phase 2 Lung Adenocarcinoma Pilot Expansion Phase Regimen A
Started | 11 | 8 | 7 | 15 | 0 | 4 | 0
Completed | 1 | 0 | 2 | 1 | 0 | 0 | 0
Not Completed | 10 | 8 | 5 | 14 | 0 | 4 | 0
Not completed — Changed treatment, too early to assess | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 1 | 0 | 2 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Developed antibodies | 7 | 2 | 3 | 8 | 0 | 0 | 0
Not completed — Refused further treatment | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Progressive disease | 1 | 2 | 2 | 3 | 0 | 2 | 0
Not completed — Treatment delay >3 weeks | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Complicating disease/intercurr. illness | 0 | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Death on study | 0 | 0 | 0 | 1 | 0 | 0 | 0
Period: Dose De-escalation of Regimen A
Arm/Group | Mesothelioma Pilot Phase Regimen A | Mesothelioma Pilot Phase Regimen B | Phase 2 Peritoneal Mesothelioma Pilot Expansion Phase | Phase 2 Pleural Mesothelioma Pilot Expansion Phase | Mesothelioma Positive Ca Dose De-escalation Pilot Regimen A | Phase 2 Pancreatic Adenocarcinoma Pilot Phase Regimen A | Phase 2 Lung Adenocarcinoma Pilot Expansion Phase Regimen A
Started | 0 | 0 | 0 | 0 | 8 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 2 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 6 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Deveoped antibodies | 0 | 0 | 0 | 0 | 3 | 0 | 0
Not completed — Progressive disease | 0 | 0 | 0 | 0 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Population: No pts were enrolled in Grp7.
Groups:
- Total: Total of all reporting groups
Arm/Group | Mesothelioma Pilot Phase Regimen A | Mesothelioma Pilot Phase Regimen B | Phase 2 Peritoneal Mesothelioma Pilot Expansion Phase | Phase 2 Pleural Mesothelioma Pilot Expansion Phase | Phase 2 Pancreatic Adenocarcinoma Pilot Phase Regimen A | Phase 2 Lung Adenocarcinoma Pilot Expansion Phase Regimen A | Total
Number analyzed (Participants) | 11 | 8 | 7 | 15 | 4 | 0 | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 9 | 7 | 6 | 7 | 4 | 0 | 33
  >=65 years | 2 | 1 | 1 | 8 | 0 | 0 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.27 (7.68) | 60.55 (16.41) | 49.91 (16.32) | 64.21 (7.65) | 52.53 (6.77) |  | 56.49 (10.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 2 | 5 | 1 |  | 14
  Male | 7 | 6 | 5 | 10 | 3 |  | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 1 | 0 |  | 1
  Not Hispanic or Latino | 11 | 8 | 7 | 14 | 4 |  | 44
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 |  | 0
  Asian | 1 | 0 | 0 | 1 | 0 |  | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 |  | 0
  Black or African American | 0 | 0 | 1 | 0 | 0 |  | 1
  White | 10 | 8 | 6 | 14 | 4 |  | 42
  More than one race | 0 | 0 | 0 | 0 | 0 |  | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 |  | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 11 | 8 | 7 | 15 | 4 |  | 45
Count of Participants with a Peritoneum and Pleural Tumor Site [Count of Participants; unit: Participants] — The peritoneum is the membrane lining the abdomen. Pleural refers to the fluid filled space between each lung.
  Participants
    Peritoneum | 2 | 1 | 7 | 0 | 0 |  | 10
    Pleural | 9 | 7 | 0 | 15 | 0 |  | 31
    Pancreatic | 0 | 0 | 0 | 0 | 4 |  | 4

OUTCOME MEASURES:

1. Primary Outcome: Response Assessment
Description: Response was assessed by the European Organization for Research and Treatment of Cancer (EORTC) modified Response Evaluation Criteria in Solid Tumors (RECIST) criteria. Complete response (CR) is complete disappearance of all target lesions. Partial response (PR) is at least a 30% decrease in the sum of the longest diameter (LD) of target lesions. Progressive disease (PD) disease is at least a 20% increase in the sum of the LD of target lesions. Stable disease (SD) is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started.
Time Frame: 52 months and 4 days
Population: No pts. were enrolled in the Phase 2 Lung Adenocarcinoma Pilot group.
Measure: Count of Participants; unit: Participants
Groups:
- Mesothelioma Pilot Phase Regimen: Drug: Pentostatin Regimen B: Cycle 1: 4 mg/m^2 or 2 mg/m^2 on days 1, 5, 9, 13 and 17 of 38 day cycle Cycles 2-6: 4 mg/m^2 on days 1 and 5 of 25 day cycle Regimen B: Cycle 1: 4 mg/m^2 on days 1, 5, 9, 13 and 17 of 38 day cycle Cycles 2-6: 4 mg/m^2 on days 1 and 5 of 25 day cycle
  Other Names:
  • Nipent Drug: Cyclophosphamide Regimen B:Cycle 1: 200 mg/day on days 1-20 of 38 day cycle Cycles 2-4: 200 mg/day on days 1-8 of 25 day cycle
  Other Names:
  • Cytoxan Drug: SS1 (dsFv)PE38 Regimen B: Cycle 1: 35mcg/kg days 18, 20, and 22. Cycles 2-4: (Days 6, 8, and 10), for a maximum of six treatment cycles.
Arm/Group | Mesothelioma Pilot Phase Regimen A | Mesothelioma Pilot Phase Regimen | Phase 2 Peritoneal Mesothelioma Pilot Expansion Phase | Phase 2 Pleural Mesothelioma Pilot Expansion Phase | Phase 2 Pancreatic Adenocarcinoma Pilot Phase Regimen A | Phase 2 Lung Adenocarcinoma Pilot Expansion Phase Regimen A
Number analyzed (Participants) | 11 | 8 | 7 | 15 | 4 | 0
Participants
  Complete Response | 0 | 0 | 0 | 0 | 0 |
  Partial Response | 2 | 0 | 0 | 0 | 0 |
  Stable Disease | 5 | 6 | 6 | 6 | 1 |
  Progressive Disease | 3 | 1 | 1 | 3 | 2 |

2. Primary Outcome: Count of Participants With SS1P Antibody Formation
Description: Development of antibodies following treatment with SS1P. The goal was to delay development of antibodies to SS1P so a patient could get a second cycle of therapy with SS1P.
Time Frame: On last day of last dosing cycle, end of cycle 1 (day 30)
Population: No pts. were enrolled in the Phase 2 Lung Adenocarcinoma Pilot group.
Measure: Count of Participants; unit: Participants
Arm/Group | Mesothelioma Pilot Phase Regimen A | Mesothelioma Pilot Phase Regimen B | Phase 2 Peritoneal Mesothelioma Pilot Expansion Phase | Phase 2 Pleural Mesothelioma Pilot Expansion Phase | Phase 2 Pancreatic Adenocarcinoma Pilot Phase Regimen A | Phase 2 Lung Adenocarcinoma Pilot Expansion Phase Regimen A
Number analyzed (Participants) | 11 | 8 | 7 | 15 | 4 | 0
Participants | 6 | 2 | 3 | 7 | 0 | 0

3. Primary Outcome: Count of Participants With Serious and Non-serious Adverse Events Assessed by the Common Terminology Criteria in Adverse Events (CTCAE v4.0) Who Were Administered SS1P and Pentostatin or Cyclophosphamide
Description: Here is the count of participants with serious and non-serious adverse events assessed by the Common Terminology Criteria in Adverse Events (CTCAE v4.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, approximately 64 months and 26 days
Population: No pts. were enrolled in the Phase 2 Lung Adenocarcinoma Pilot group.
Measure: Count of Participants; unit: Participants
Arm/Group | Mesothelioma Pilot Phase Regimen A | Mesothelioma Pilot Phase Regimen B | Phase 2 Peritoneal Mesothelioma Pilot Expansion Phase | Phase 2 Pleural Mesothelioma Pilot Expansion Phase | Phase 2 Pancreatic Adenocarcinoma Pilot Phase Regimen A | Phase 2 Lung Adenocarcinoma Pilot Expansion Phase Regimen A
Number analyzed (Participants) | 11 | 8 | 7 | 15 | 4 | 0
Participants | 11 | 8 | 7 | 15 | 4 | 0

4. Primary Outcome: Recommended Phase 2 Dose (RP2D) in Drug Lot FIL129J01
Description: Should any 2 patients within the first 3 to 6 patients experience treatment limiting toxicity requiring cessation of treatment prior to the conclusion of the first cycle, the maximum tolerated dose will have been exceeded and patients will be enrolled to the next lower dose.
Time Frame: Days 1, 3, and 5 of a 21 day cycle
Measure: Number; unit: mcg/kg/dose
Groups:
- Meso., Peritoneal, Pleural & Pancreatic Regimen A: Drug: Pentostatin Regimen A: Cycle 1: 4 mg/m^2 on days 1, 5 and 9 of 30 day cycle Cycles 2-4: 4 mg/m^2 on day 1 of 21 day cycle
  Other Names:
  • Nipent Drug: Cyclophosphamide Regimen A:Cycle 1: 200 mg/day on days 1-12 of 30 day cycle Cycles 2-4: 200 mg/day on days 1-4 of 21 day cycle
  Other Names:
  • Cytoxan
  Drug: SS1(dsFv)PE38 Regimen A: Cycle 1: 35 mcg/kg or 25 mcg/kg days 10, 12 and 14. Cycles 2-4: Days 2, 4, and 6, for a maximum of six treatment cycles.
  During Phase 2 SS1P was administered from 2 different Lots at 35mcg/kg (Lot F1L129J01 and Lot07310809). It was discovered that Lot F1L129J01 was more potent than Lot 07310809, therefore, a dose de-escalation was done for 8 participants who received that Lot to determine the MTD specific to the Lot.
Arm/Group | Meso., Peritoneal, Pleural & Pancreatic Regimen A
Number analyzed (Participants) | 8
mcg/kg/dose | 25

5. Secondary Outcome: Overall Survival
Description: The Kaplan-Meier was used to determine the probability of overall survival from on-study date until death or last follow-up (calculated from the date of study entry until the date of analysis).
Time Frame: 36 months
Population: No pts. were enrolled in the Phase 2 Lung Adenocarcinoma Pilot group.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Mesothelioma Pilot Phase Regimen A | Mesothelioma Pilot Phase Regimen B | Phase 2 Peritoneal Mesothelioma Pilot Expansion Phase | Phase 2 Pleural Mesothelioma Pilot Expansion Phase | Phase 2 Pancreatic Adenocarcinoma Pilot Phase Regimen A | Phase 2 Lung Adenocarcinoma Pilot Expansion Phase Regimen A
Number analyzed (Participants) | 11 | 8 | 7 | 15 | 4 | 0
Months | 8.9 [5.4 to 32.2] | 11.2 [1.0 to 13.0] | 29.3 [3.4 to 29.3] | 4.2 [2.0 to 7.9] | 9.3 [1.2 to 15.1] |

6. Secondary Outcome: Progression-free Survival
Description: Defined as the time interval from the start of treatment to documented evidence of disease progression. Progressive disease is assessed by the European Organization for Research and Treatment of Cancer (EORTC) modified Response Evaluation Criteria in Solid Tumors (RECIST) criteria, and is at least a 20% increase in the sum of the longest diameter (LD) of target lesions, taking as reference the smallest sum on study LD (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5mm. (Note: the appearance of one or more new lesions is also considered progression).
Time Frame: 36 months
Population: No pts. were enrolled in the Phase 2 Lung Adenocarcinoma Pilot group.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Meothelioma Pilot Phase Phase Regimen A: Drug: Pentostatin Regimen A: Cycle 1: 4 mg/m^2 on days 1, 5 and 9 of 30 day cycle Cycles 2-4: 4 mg/m^2 on day 1 of 21 day cycle
  Other Names:
  • Nipent Drug: Cyclophosphamide Regimen A:Cycle 1: 200 mg/day on days 1-12 of 30 day cycle Cycles 2-4: 200 mg/day on days 1-4 of 21 day cycle
  Other Names:
  • Cytoxan Drug: SS1 (dsFv)PE38 Regimen A: Cycle 1: 35 mcg/kg days 10, 12, and 14. Cycles 2-4: Days 2, 4, and 6, for a maximum of six treatment cycles
- Meothelioma Pilot Phase Regimen B: Drug: Pentostatin Regimen B: Cycle 1: 4 mg/m^2 or 2 mg/m^2 on days 1, 5, 9, 13 and 17 of 38 day cycle Cycles 2-6: 4 mg/m^2 on days 1 and 5 of 25 day cycle Regimen B: Cycle 1: 4 mg/m^2 on days 1, 5, 9, 13 and 17 of 38 day cycle Cycles 2-6: 4 mg/m^2 on days 1 and 5 of 25 day cycle
  Other Names:
  • Nipent Drug: Cyclophosphamide Regimen B:Cycle 1: 200 mg/day on days 1-20 of 38 day cycle Cycles 2-4: 200 mg/day on days 1-8 of 25 day cycle
  Other Names:
  • Cytoxan Drug: SS1 (dsFv)PE38 Regimen B: Cycle 1: 35mcg/kg days 18, 20, and 22. Cycles 2-4: (Days 6, 8, and 10), for a maximum of six treatment cycles.
Arm/Group | Meothelioma Pilot Phase Phase Regimen A | Meothelioma Pilot Phase Regimen B | Phase 2 Peritoneal Mesothelioma Pilot Expansion Phase | Phase 2 Pleural Mesothelioma Pilot Expansion Phase | Phase 2 Pancreatic Adenocarcinoma Pilot Phase Regimen A | Phase 2 Lung Adenocarcinoma Pilot Expansion Phase Regimen A
Number analyzed (Participants) | 11 | 8 | 7 | 15 | 4 | 0
Months | 11.8 [1.6 to 13.6] | 8.8 [0.6 to 13.0] | 8.9 [1.8 to NA] — Upper bound confidence interval is undefined because there are too few subjects and progressions after the median time to estimate the confidence bound; it cannot be calculated. | 3.9 [1.6 to 6.4] | 4.4 [0.9 to 7.4] |

7. Secondary Outcome: Duration of Response
Description: DOR is assessed by the European Organization for Research and Treatment of Cancer (EORTC) modified Response Evaluation Criteria in Solid Tumors (RECIST) criteria and is measured from the time measurement criteria is met for complete response or partial response (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented (taking as reference for progressive disease the smallest measurements recorded since the treatment started). Complete response is disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to<10mm. partial response is at least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD. Progressive disease is at least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum on study LD (this includes the baseline sum if that is the smallest on study).
Time Frame: up to 2.5 years
Population: In months; the only 3 responders were in group one, thus arm/groups 2-7 are not shown here.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Mesothelioma Pilot Phase Regimen A
Number analyzed (Participants) | 3
Months | 16.3 [10.6 to 26.2]

8. Other Pre Specified Outcome: Count of Participants SS1P Cycles Received Following Onstudy
Description: Here are the number of participants who had SS1P cycles during cycle 1-6.
Time Frame: Cycles 1-6, up to 180 days
Population: No pts. were enrolled in the Phase 2 Lung Adenocarcinoma Pilot group.
Measure: Count of Participants; unit: Participants
Arm/Group | Mesothelioma Pilot Phase Regimen A | Mesothelioma Pilot Phase Regimen B | Phase 2 Peritoneal Mesothelioma Pilot Expansion Phase | Phase 2 Pleural Mesothelioma Pilot Expansion Phase | Phase 2 Pancreatic Adenocarcinoma Pilot Phase Regimen A | Phase 2 Lung Adenocarcinoma Pilot Expansion Phase Regimen A
Number analyzed (Participants) | 11 | 8 | 7 | 15 | 4 | 0
Participants
  SS1P 1 Cycle | 1 | 3 | 0 | 5 | 2 | 0
  SS1P 2 Cycles | 8 | 0 | 4 | 8 | 1 | 0
  SS1P 3 Cycles | 0 | 3 | 0 | 1 | 1 | 0
  SS1P 4 Cycles | 1 | 1 | 3 | 0 | 0 | 0
  SS1P 5 Cycles | 0 | 1 | 0 | 1 | 0 | 0
  SS1P 6 Cycles | 1 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 64 months and 26 days.
Description: No pts. were enrolled in the Phase 2 Lung Adenocarcinoma Pilot group.
Groups:
- Mesothelioma Positive Ca Dose De-escalation Pilot Regimen A: Drug: Pentostatin Regimen A: Cycle 1: 4 mg/m^2 on days 1, 5 and 9 of 30 day cycle Cycles 2-4: 4 mg/m^2 on day 1 of 21 day cycle
  Other Names:
  • Nipent Drug: Cyclophosphamide Regimen A:Cycle 1: 200 mg/day on days 1-12 of 30 day cycle Cycles 2-4: 200 mg/day on days 1-4 of 21 day cycle
  Other Names:
  • Cytoxan Drug: SS1(dsFv)PE38 Regimen A: Cycle 1: 35 mcg/kg or 25 mcg/kg days 10, 12 and 14. Cycles 2-4: Days 2, 4, and 6, for a maximum of six treatment cycles
  During Phase 2 SS1P was administered from 2 different Lots at 35mcg/kg (Lot F1L129J01 and Lot07310809). It was discovered that Lot F1L129J01 was more potent than Lot 07310809, therefore, a dose de-escalation was done for 8 participants who received that Lot to determine the MTD specific to the Lot.
Arm/Group | Mesothelioma Pilot Phase Regimen A | Mesothelioma Pilot Phase Regimen B | Phase 2 Peritoneal Mesothelioma Pilot Expansion Phase | Phase 2 Pleural Mesothelioma Pilot Expansion Phase | Mesothelioma Positive Ca Dose De-escalation Pilot Regimen A | Phase 2 Pancreatic Adenocarcinoma Pilot Phase Regimen A | Phase 2 Lung Adenocarcinoma Pilot Expansion Phase Regimen A
All-Cause Mortality (participants affected / at risk) | 5/11 | 8/8 | 3/7 | 9/15 | 1/8 | 1/4 | 0/0
Serious Adverse Events (participants affected / at risk) | 6/11 | 8/8 | 3/7 | 9/15 | 1/8 | 1/4 | 0/0
Other Adverse Events (participants affected / at risk) | 11/11 | 8/8 | 7/7 | 15/15 | 8/8 | 4/4 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mesothelioma Pilot Phase Regimen A (N=11) | Mesothelioma Pilot Phase Regimen B (N=8) | Phase 2 Peritoneal Mesothelioma Pilot Expansion Phase (N=7) | Phase 2 Pleural Mesothelioma Pilot Expansion Phase (N=15) | Mesothelioma Positive Ca Dose De-escalation Pilot Regimen A (N=8) | Phase 2 Pancreatic Adenocarcinoma Pilot Phase Regimen A (N=4) | Phase 2 Lung Adenocarcinoma Pilot Expansion Phase Regimen A (N=0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Death NOS (General disorders) | 5 (5) | 5 (5) | 2 (2) | 4 (4) | 0 (0) | 1 (1) | 0 (0)
Fever (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 | 0 (0) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3) | 1 (1) | 4 (4) | 1 (1) | 0 (0) | 0 (0) — Death
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Death
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mesothelioma Pilot Phase Regimen A (N=11) | Mesothelioma Pilot Phase Regimen B (N=8) | Phase 2 Peritoneal Mesothelioma Pilot Expansion Phase (N=7) | Phase 2 Pleural Mesothelioma Pilot Expansion Phase (N=15) | Mesothelioma Positive Ca Dose De-escalation Pilot Regimen A (N=8) | Phase 2 Pancreatic Adenocarcinoma Pilot Phase Regimen A (N=4) | Phase 2 Lung Adenocarcinoma Pilot Expansion Phase Regimen A (N=0)
Activated partial thromboplastin time prolonged (Investigations) | 2 (2) | 5 (10) | 1 (2) | 7 (10) | 3 (6) | 2 (5) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 2 (4) | 2 (6) | 2 (2) | 2 (4) | 1 (1) | 0 (0)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 6 (17) | 4 (15) | 2 (2) | 7 (19) | 5 (10) | 4 (7) | 0 (0)
Alkaline phosphatase increased (Investigations) | 2 (4) | 3 (13) | 3 (10) | 3 (5) | 3 (11) | 2 (5) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 8 (31) | 7 (44) | 4 (28) | 11 (39) | 8 (35) | 4 (12) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 6 (7) | 3 (3) | 3 (5) | 3 (3) | 2 (4) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (2) | 2 (2) | 2 (3) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Injury, poisoning and procedural complications) | 7 (20) | 4 (17) | 3 (12) | 7 (19) | 6 (16) | 4 (9) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Asystole (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 2 (3) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Atrial flutter (Cardiac disorders) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (6) | 0 (0) | 1 (4) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Bloating (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 2 (4) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blurred vision (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Capillary leak syndrome (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac disorders - Other, (coronary artery disease) (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Chills (General disorders) | 1 (1) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusion (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 8 (12) | 2 (3) | 4 (7) | 6 (10) | 7 (9) | 4 (4) | 0 (0)
Corneal ulcer (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 5 (5) | 2 (2) | 1 (1) | 0 (0)
Creatinine increased (Investigations) | 3 (7) | 3 (14) | 2 (4) | 7 (12) | 4 (8) | 2 (5) | 0 (0)
Dehydration (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 2 (2) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 5 (5) | 4 (8) | 3 (5) | 5 (9) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 3 (4) | 6 (8) | 3 (3) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Edema face (General disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Edema limbs (General disorders) | 6 (10) | 5 (9) | 3 (6) | 11 (29) | 5 (10) | 2 (2) | 0 (0)
Ejection fraction decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Erythroderma (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 7 (11) | 4 (11) | 4 (8) | 9 (11) | 7 (11) | 4 (5) | 0 (0)
Fever (General disorders) | 1 (3) | 4 (15) | 1 (1) | 8 (10) | 4 (8) | 2 (6) | 0 (0)
Flashing lights (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 2 (2) | 1 (1) | 3 (4) | 2 (2) | 1 (1) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hot flashes (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 2 (6) | 2 (8) | 4 (7) | 0 (0) | 0 (0) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 10 (35) | 6 (28) | 5 (12) | 15 (71) | 6 (20) | 2 (11) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 3 (10) | 2 (12) | 5 (12) | 7 (13) | 4 (7) | 1 (1) | 0 (0)
Hypermagnesemia (Metabolism and nutrition disorders) | 5 (7) | 4 (7) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (3) | 2 (2) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 3 (19) | 3 (5) | 6 (14) | 3 (6) | 0 (0) | 0 (0)
Hyperuricemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (8) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 11 (34) | 7 (57) | 6 (38) | 12 (66) | 8 (37) | 4 (13) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (2) | 1 (10) | 1 (5) | 7 (17) | 3 (10) | 1 (6) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 1 (1) | 2 (5) | 1 (1) | 1 (1) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 5 (7) | 4 (21) | 2 (3) | 5 (13) | 1 (1) | 0 (0) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 8 (26) | 5 (11) | 7 (22) | 13 (45) | 8 (28) | 4 (11) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (5) | 4 (23) | 4 (6) | 9 (37) | 4 (8) | 2 (3) | 0 (0)
Hypotension (Vascular disorders) | 2 (2) | 3 (5) | 1 (2) | 8 (13) | 3 (4) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (4) | 1 (2) | 5 (9) | 1 (1) | 0 (0) | 0 (0)
Infections and infestations - Other, (folliculitis on abdomen and back) (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 3 (3) | 1 (1) | 2 (2) | 6 (7) | 2 (3) | 1 (1) | 0 (0)
Laryngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 11 (121) | 8 (86) | 7 (83) | 15 (140) | 8 (84) | 4 (22) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, (muscle twitching) (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 8 (9) | 5 (7) | 5 (12) | 13 (28) | 7 (10) | 2 (2) | 0 (0)
Nervous system disorders - Other, (vocal cord paralysis) (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 2 (4) | 5 (16) | 1 (3) | 3 (9) | 3 (13) | 2 (10) | 0 (0)
Non-cardiac chest pain (Musculoskeletal and connective tissue disorders) | 5 (8) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (2) | 4 (7) | 2 (2) | 1 (1) | 0 (0)
Paresthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 3 (11) | 7 (29) | 2 (4) | 4 (6) | 3 (7) | 2 (4) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Photophobia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 2 (2) | 5 (12) | 1 (2) | 0 (0) | 0 (0)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other, (tachypnea) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Restlessness (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 2 (2) | 0 (0) | 4 (5) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 3 (3) | 2 (3) | 5 (10) | 3 (4) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Rash, face, upper torso
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Superior vena cava syndrome (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (6) | 1 (2) | 0 (0) | 0 (0)
Thromboembolic event (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 3 (7) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Vasovagal reaction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ventricular arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (4) | 3 (6) | 4 (8) | 6 (16) | 3 (4) | 1 (1) | 0 (0)
Weight gain (Investigations) | 4 (6) | 3 (4) | 2 (4) | 8 (25) | 2 (3) | 0 (0) | 0 (0)
Weight loss (Investigations) | 0 (0) | 1 (4) | 2 (4) | 2 (7) | 2 (4) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
White blood cell decreased (Investigations) | 8 (33) | 7 (70) | 5 (25) | 11 (55) | 7 (36) | 3 (19) | 0 (0)
Infections and infestations - Other, (tinea corporis on nape of neck) (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2017-07-06): https://cdn.clinicaltrials.gov/large-docs/90/NCT01362790/Prot_SAP_ICF_000.pdf